CLINICAL TRIAL: NCT06138184
Title: Patient Education for Anticoagulants Using Learning Theories - a Pilot Study
Brief Title: Learning Theory Patient Education for Anticoagulants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Aubrey E. Jones, Assistant Research Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB_00146488; K23HL157751 (NIH)
Record Dates: First submitted 2022-12-16; First posted 2023-11-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: anticoagulant; direct oral anticoagulant; vitamin k antagonist; warfarin; patient education; learning theory
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard Educational process
  Interventions: Behavioral: Control Group: Standard of Care
- Education Intervention (Experimental): New educational intervention
  Interventions: Behavioral: Anticoagulation Educational Materials

INTERVENTIONS:
Behavioral: Anticoagulation Educational Materials — This includes new web-based patient educational materials that have been developed prior to the start of the study
  Arms: Education Intervention
Behavioral: Control Group: Standard of Care — This will be the current practice for patient education
  Arms: Standard Care

SUMMARY:
The goal of this study is to test the feasibility of a randomized control trial evaluating the educational tool for anticoagulated patients.

Participants will be randomized to use new educational materials or current existing educational materials and answer survey questions.

DETAILED DESCRIPTION:
Eligible patients will be randomized using stratified block randomization to control for the type of anticoagulant (warfarin vs. DOAC) and status (naïve vs. experienced) to either the education intervention from Aim 2 or standard of care Data will be collected via online surveys before the intervention, immediately after, and then 3 months after the intervention.

Patients at the University of Utah Thrombosis Clinic will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* initiating (naïve) or currently taking (experienced) oral anticoagulants with an anticipated treatment duration of at least three months
* Experienced patients will be eligible if they score less than 75% on the Anticoagulation Knowledge Test

Exclusion Criteria:

* Deficits in cognitive abilities, sensory input, or language significant enough to impede their use of the education tool and/or provision of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing a randomized control trial | 18 months
  The study will be feasible if 1) the consent rate if 5 patients per month, 2) Proportion of patients completing the educational tool is 90%; 3) Loss to follow-up at three months is 20% or less

SECONDARY OUTCOMES:
Acceptability | 3 months
  High acceptability based on self-reported questionnaires using Likert questions per the Theoretical Framework of Acceptability domains
Acceptability - Educational Tool | At time of intervention
  This will be measured using an adapted version of the Ottawa Decision Aid Acceptability Measures which is a 10-question tool shortened to 5 questions that assess: 1) The way information is presented, 2) Length of the Materials, 3) Amount of information, 4) What was liked, and 5) Suggestions for improvement
Acceptability - Workflow Disruption | 18 months
  2 questions to providers asking to rate how much a) the study disrupted their workflow and b) how much the educational tool disrupted their workflow on a scale from 1- Very disruptive to 5 - Not all disruptive. Higher scores are better outcomes
Acceptability - Satisfaction | 3 months
  Patients and providers will both complete a 5 point Likert scale asking how satisfied they are with the educational materials, with 1 being Very dissatisfied and 5 being Very Satisfied.
Acceptability - Intervention/Survey Fatigue | 3 months
  1 question measuring survey fatigue: 1) the length of surveys was a) too long, b) too short, c) just right and the number of surveys that were not filled out/not completed. If the majority of surveys are not completed or started, and the majority of patients answer that the length of surveys was too long, that will indicate high survey fatigue

OTHER OUTCOMES:
Patient knowledge | 3 months
  Anticoagulation Knowledge Test 28 item scale for patients taking warfarin or a direct oral anticoagulant to assess their knowledge , Minimum score = 0, Max score = 28. Higher scores indicate more knowledge
Information overload | 3 months
  adapted Cancer Information Overload Scale 5-item scale from Strongly Disagree to Strongly Agree. Minimum score = 5, maximum score = 20. The higher the score indicates higher information overload.
Adherence | 3 months
  Visual Analog Rating Scale (VAS) asks patients to estimate in a specified time period (the 3 months of the study period), the percentage of medication doses that they have taken as prescribed (0-100%) Higher percentage means higher adherence.
Clinical outcomes | 3 months
  Patients will report the number (if any) of thromboembolic (stroke, deep vein thrombosis, pulmonary or systemic embolism), or bleeding events that they have had during the study period. We will also review patient charts to see if there are any reported events in the chart that are not reported by the patient. Bleeding events will be classified into major or clinically relevant non-major bleeding according to the International Society on Thrombosis and Haemostasis (ISTH) definitions. We will also monitor for any deaths that may occur.

CONTACTS AND LOCATIONS:
Overall Officials: Aubrey E Jones, PharmD, MSCI, Principal Investigator — University of Utah